CLINICAL TRIAL: NCT02461342
Title: Genetic, Environment and Its Interaction Analysis for Cardiovascular Autonomic Neuropathy in Chinese Population
Brief Title: Genetic, Environment and Its Interaction Analysis for Cardiovascular Autonomic Neuropathy
Status: Completed | Type: Observational
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Collaborators: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Zihui Tang, M.D and Ph.D, Huashan Hospital
Other Study IDs: CANGEI_Dr.Tang
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Cardiovascular Autonomic Neuropathy
Keywords: Genetic; environment; interaction analysis; cardiovascular autonomic neuropathy; CAN

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNAs were extracted and genetyped by using SNP.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dr.Tang's research group: Dr.Tang's research group for genetic, environment and its interaction analysis of human complex disease
  Interventions: Other: not intervention

INTERVENTIONS:
Other: not intervention — This is a cross-sectional study, no intervention was performed.
  Other Names: nothing

SUMMARY:
A large-scale, community-based, cross-sectional study was conducted to explore the extent to which genetic, environment and its interactions associated with cardiovascular autonomic neuropathy (CAN) in general Chinese population. A total of more than 2000 participants were recruited by using multiple stages sampling (first cluster sampling and then simply sampling). Data involved in variables of genetic, environment were collected. Every participants was complete DNA extracted and genotyped by using single nucleotide polymorphism (SNP). Cardiovascular autonomic functions were measured by using short-term heart rate variability (HRV) to evaluate the outcome of CAN. Genetic analysis were employed to evaluate genetic variants, environmental risk factors and its interactions for CAN.

DETAILED DESCRIPTION:
A large-scale, community-based, cross-sectional study was conducted to explore the extent to which genetic, environment and its interactions associated with cardiovascular autonomic neuropathy (CAN) in general Chinese population. A total of more than 2000 participants were recruited by using multiple stages sampling (first cluster sampling and then simply sampling). Data involved in variables of genetic, environment were collected. Every participant was complete DNA extracted and genotyped by using single nucleotide polymorphism (SNP). Cardiovascular autonomic functions were measured by using short-term heart rate variability (HRV) to evaluate the outcome of CAN. Genetic analysis were employed to evaluate genetic variants, environmental risk factors and its interactions for CAN.Univariate and multiple variables analysis have been performed to examine potential environmental and genetic risk factors of CAN.

ELIGIBILITY:
Inclusion Criteria:

* Survey Chinese participants with undiagnosed CAN Aged 30-90 years, were included in this study.

Exclusion Criteria:

-

Some subjects were excluded from the study to eliminate potential confounding factors that may have influenced their CA function. Briefly, the exclusion criteria were as follows:

1. history or findings of arrhythmia and hyperthyroidism or hypothyroidism
2. pregnancy or lactation
3. serious hepatic or renal dysfunctions (GFR < 30 mL/min/1.73m2). Of these subjects, complete baseline data were obtained for 2,092 (69.46%) of the participants.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators recruited participants from rural and urban communities in Shanghai. Survey participants with undiagnosed CAN, aged 30-90 years, were included in this study. Our study invited a total of 3,012 subjects to a screening visit between 2011 and 2012.
Sampling Method: Probability Sample
Enrollment: 2100 (Actual)
Dates: Start 2011-01; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
cardiovascular autonomic neuropathy (CAN) measured by short-term heart rate variability (HRV) | participants will be measured for the duration of outpatient stay, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zihui Tang, M.D and Ph.D, Principal Investigator — Huashan Hospital
Locations (2):
- China (2):
  - Huasha Hospital, Shanghai, Shanghai Municipality
  - Huashan Hospital, Shanghai, Shanghai Municipality

REFERENCES:
- [Result] Liao XP, Zhu HW, Zeng F, Tang ZH. The association and interaction analysis of hypertension and uric acid on cardiovascular autonomic neuropathy. J Endocrinol Invest. 2015 Oct;38(10):1075-82. doi: 10.1007/s40618-015-0291-x. Epub 2015 Apr 23. PMID 25903694
- [Result] Tang ZH, Zeng F, Zhang XZ. Human genetics of diabetic nephropathy. Ren Fail. 2015 Apr;37(3):363-71. doi: 10.3109/0886022X.2014.1000801. Epub 2015 Jan 16. PMID 25594612
- [Result] Zhang L, Tang ZH, Zeng F, Li Z, Zhou L, Li Y. Clinical risk model assessment for cardiovascular autonomic dysfunction in the general Chinese population. J Endocrinol Invest. 2015 Jun;38(6):615-22. doi: 10.1007/s40618-014-0229-8. Epub 2015 Jan 3. PMID 25555369
- [Result] Tang ZH, Wang L, Zeng F, Li Z, Yu X, Zhang K, Zhou L. Bayesian estimation of cardiovascular autonomic neuropathy diagnostic test based on short-term heart rate variability without a gold standard. BMJ Open. 2014 Oct 6;4(9):e005096. doi: 10.1136/bmjopen-2014-005096. PMID 25287103
- [Result] Tang ZH, Wang L, Zeng F, Zhang K. Human genetics of diabetic retinopathy. J Endocrinol Invest. 2014 Dec;37(12):1165-74. doi: 10.1007/s40618-014-0172-8. Epub 2014 Sep 9. PMID 25201002
- [Result] Tang ZH, Zeng F, Li Z, Zhou L. Association and predictive value analysis for resting heart rate and diabetes mellitus on cardiovascular autonomic neuropathy in general population. J Diabetes Res. 2014;2014:215473. doi: 10.1155/2014/215473. Epub 2014 Mar 18. PMID 24772443
- [Result] Zeng F, Tang ZH, Li Z, Yu X, Zhou L. Normative reference of short-term heart rate variability and estimation of cardiovascular autonomic neuropathy prevalence in Chinese people. J Endocrinol Invest. 2014 Apr;37(4):385-91. doi: 10.1007/s40618-013-0047-4. Epub 2014 Jan 9. PMID 24633734
- [Result] Tang ZH, Zeng F, Yu X, Zhou L. Bayesian estimation of cardiovascular autonomic neuropathy diagnostic test based on baroreflex sensitivity in the absence of a gold standard. Int J Cardiol. 2014 Feb 15;171(3):e78-80. doi: 10.1016/j.ijcard.2013.11.100. Epub 2013 Dec 6. No abstract available. PMID 24360155
- [Result] Tang ZH, Liu J, Zeng F, Li Z, Yu X, Zhou L. Comparison of prediction model for cardiovascular autonomic dysfunction using artificial neural network and logistic regression analysis. PLoS One. 2013 Aug 5;8(8):e70571. doi: 10.1371/journal.pone.0070571. Print 2013. PMID 23940593
- [Result] Tang ZH, Zeng F, Li Z, Zhou L. A risk score of cardiovascular autonomic dysfunction for targeted screening in the Chinese population. Int J Cardiol. 2013 Oct 12;168(5):4861-2. doi: 10.1016/j.ijcard.2013.07.062. Epub 2013 Jul 25. No abstract available. PMID 23890865
- [Result] Li Z, Tang ZH, Zeng F, Zhou L. Associations between the severity of metabolic syndrome and cardiovascular autonomic function in a Chinese population. J Endocrinol Invest. 2013 Dec;36(11):993-9. doi: 10.3275/9005. Epub 2013 Jun 17. PMID 23770583
- [Result] Tang ZH, Fang Z, Zhou L. Human genetics of diabetic vascular complications. J Genet. 2013 Dec;92(3):677-94. doi: 10.1007/s12041-013-0288-1. PMID 24371189
- [Derived] Lv Y, Zhou L, Tang Z, Dong J. Association and interaction analysis of diabetes mellitus and SCN10A for cardiovascular autonomic neuropathy in a Chinese population. Postgrad Med J. 2017 Jun;93(1100):344-348. doi: 10.1136/postgradmedj-2016-134202. Epub 2016 Oct 11. PMID 27729462
- [Derived] Zeng F, Zhou L, Tang Z. A study for association and interaction analysis to metabolic syndrome and the ESR1 gene on cardiovascular autonomic neuropathy in a Chinese Han population. Diabetol Metab Syndr. 2016 Jul 22;8:42. doi: 10.1186/s13098-016-0155-3. eCollection 2016. PMID 27453734